CLINICAL TRIAL: NCT00922090
Title: A Non-interventional Study Evaluating the Clinical Benefit and Effectiveness of Quetiapine Fumarate Extended-Release Tablets (SEROQUEL XRâ) in Subjects With Schizophrenia-An Observational, Multicentric Prospective Study
Brief Title: A Non-interventional Study Evaluating the Clinical Benefit and Effectiveness of Quetiapine Fumarate Extended
Acronym: CLIMAX
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Korea
Other Study IDs: NIS-NKR-SER-2009/1
Record Dates: First submitted 2009-06-12; First posted 2009-06-17 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Seroquel XR; CGI-CB; SWN-K
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this NIS is to assess the clinical benefit subjects derive from taking seroquel XR, using the CGI-CB. The secondary objective is to assess the effectiveness,safety and tolerability of seroquel XR tablets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Schizophrenia according to DSM-IV-TR criteria
* Patients who are taking Seroquel XR no longer than 1 month
* Patients who get antipsychotics monotherapy at least 1 week before enroll in this study

Exclusion Criteria:

* First episode, drug naive schizophrenic subjects.
* Meeting the criteria for any other (than schizophrenia) DSM-IV Axis I diagnosis,concomitant organic mental disorder or mental retardation that in the opinion of the Principal Investigator may interfere with study conduct or interpretation.
* Known lack of response to clozapine or treatment with clozapine within 4 weeks prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diagnosed as Schizophrenia according to DSM-IV-TR criteria, the groups will be selected selected from general hospital or mental hospital.
Sampling Method: Probability Sample
Enrollment: 1494 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the Clinical Global Impression score - Clinical Benefit Scale (CGI-CB) after 2 months of treatment with Seroquel XR | 8 weeks

SECONDARY OUTCOMES:
CGI-I score's change from 7th day to 8weeks | 8 weeks
Patients' ratio who've been improved CGI-S score more than 4, from baseline to 8weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JoonWoo Bahn, MD, PhD, Study Director — AstraZeneca Korea
Locations (11):
- South Korea (11):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Jeju City
  - Research Site, Kyung Gi
  - Research Site, Kyungju
  - Research Site, Kyungnam
  - Research Site, Namyangju
  - Research Site, Seoul